CLINICAL TRIAL: NCT02379039
Title: Multimodal Monitoring of Radiotherapy Response in Squamous Cell Cancer in Head & Neck, Lung, Oesophagus, Anal Canal and Uterine Cervix - a Basis for Personalised Radiotherapy
Brief Title: Multimodal Monitoring of Radiotherapy Response in Squamous Cell Cancer
Acronym: MORRIS
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: MORRIS_1
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Squamous Carcinoma; Head and Neck Cancer; Anal Cancer; Lung Cancer; Esophageal Cancer; Cervix Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Anus Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour biopsies, plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study's aim is to define imaging and molecular bio-markers for prediction of radiotherapy response of squamous cell carcinomas, in an early treatment phase.

DETAILED DESCRIPTION:
Patients with squamous cell carcinoma of the head & neck, anal canal, cervix, esophagus or lung will be assessed before start of radiotherapy and 1-2 weeks after start. Multi-parametric MRI and 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) will be performed in parallel to metabolomic analyses of tumour tissue. The investigators will correlate changes in imaging bio-markers to corresponding changes in tissue or blood bio-markers by repeated imaging and biopsies for better understanding of the image parameters.

The data from the two assessments will be used for identifying imaging bio-markers, predictive for outcome. The patient data will be divided into one set of data for hypothesis generation and another set for validation.

ELIGIBILITY:
Inclusion Criteria:

1. Morphologically (pathology or cytology) verified, previously untreated squamous cell carcinoma (SCC) of the oral cavity, oropharynx, uterine cervix, oesophagus or lung.
2. The patient should be planned for treatment with radiotherapy alone or in combination with concomitant medical therapy
3. The tumour shall be radiologically and/or visually identifiable and accessible for biopsy without the need for general anaesthesia or other major interventions
4. The patient must be at least 18 years of age, able to understand the given information and, leave a written informed consent to participate

Exclusion Criteria:

1. The patient is unwilling to participate in the study
2. Patients with adjuvant post-operative radiotherapy (i.e. no visible remaining tumour)
3. Pregnancy or lactation
4. Contraindications to investigations with MRI, gadolinium contrast or PET-tracers
5. Patients with an estimated glomerular filtration rate (GFR) <60 ml/min/1.73m2.
6. Severe co-morbidities that are judged to significantly compromise survival in a two-years perspective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously untreated squamous carcinoma aimed for radiotherapy with curative intent of the oral cavity, oropharynx, uterine cervix, oesophagus, anal canal or lung.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2015-05; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Loco regional control | 2 years
  After completion of radiotherapy

SECONDARY OUTCOMES:
Loco regional tumour control (response) | 2 months
  After completion of radiotherapy
Patterns of failure | 2 years
  Time and location of recurrence
Overall survival | 5 years
  After completion of radiotherapy
Changes in imaging and metabolic data | 1-2 weeks
  As measured 1-2 weeks after start of radiotherapy
Site specific toxicity | 1 year
  Measured as patient reported side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Björn Zackrisson, Professor, Principal Investigator — Umeå University, Department of Radiation Sciences - Oncology
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
If relevant, anonymized data may be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available 6 months after publication
Access Criteria: Metaanalysis, comprehensive review. Request is sent to principal investigator (Bjorn Zackrisson)

REFERENCES:
- [Derived] Strandberg S, Jonsson J, Zarei M, Aglund K, Blomqvist L, Soderkvist K. Baseline and early response 2-[18F]FDG-PET/MRI for prediction of radiotherapy outcome in uterine cervical squamous cell carcinoma: a prospective single-center observational cohort study. EJNMMI Rep. 2024 Mar 1;8(1):5. doi: 10.1186/s41824-024-00188-7. PMID 38748271

DOCUMENTS (1):
  • Study Protocol (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT02379039/Prot_001.pdf